CLINICAL TRIAL: NCT05521841
Title: Comparison Of Erector Spinae Plane Block With Transversus Abdominis Plane Block For Postoperative Pain Management In Patients Undergoing Total Abdominal Hysterectomy: A Randomized Controlled Trial
Brief Title: Comparison Of Erector Spinae Plane Block With Transversus Abdominis Plane Block For Postoperative Pain Management In Patients Undergoing Total Abdominal Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Dr Biplov Neupane, Resident, Department of Anesthesiology, Tribhuvan University Teaching Hospital, Institute Of Medicine., Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 92(6-11)F2
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Postoperative analgesia; ESP block; TAP block; TAH
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: hospital based randomized, prospective, interventional study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): Bilateral Ultrasound Guided Erector Spinae Plane Block
  Interventions: Procedure: Erector Spinae Plane Block(Bilateral Ultrasound Guided Erector Spinae Plane Block)
- Transversus abdominis plane block (Active Comparator): Bilateral Ultrasound-guided bilateral Transversus abdominis plane block
  Interventions: Procedure: Transversus abdominis plane block(Bilateral Ultrasound-guided bilateral Transversus abdominis plane block)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block(Bilateral Ultrasound Guided Erector Spinae Plane Block) — Bilateral USG guided Erector Spinae Plane Block:
  Drug used 20 ml of 0.25% Bupivacaine in each side. Total 40 ml volume. Dosage 100mg Ultrasound transducer will be placed in a cephalocaudal orientation over the back at 10th thoracic vertebral level.
  The probe will then slowly be moved laterally until the transverse process is visible The trapezius muscle and erector spinae muscle will be identified as superficial to the transverse process.
  A 25-gauge Quincke spinal needle (Romsons spinal needle, Quincke type)will be inserted using an in-plane approach in the cephalad to the caudal direction and towards the transverse process.
  A 5ml bolus of local anesthetic will be given. Erector spinae muscle plane is then visualized separating from the transverse process.
  The local anesthetic is then injected in 5 ml increments, with aspiration after every 5 ml to avoid intravascular injection Same procedure will be repeated on the other side
  Other Names: ESP
  Arms: Erector Spinae Plane Block
Procedure: Transversus abdominis plane block(Bilateral Ultrasound-guided bilateral Transversus abdominis plane block) — Bilateral Ultrasound-guided bilateral Transversus abdominis plane block Drug used 20 ml of 0.25% Bupivacaine in each side. Total 40 ml volume. Dosage 100mg The linear transducer will be placed in the transverse plane at the lateral abdominal wall in the mid-axillary line, between the lower costal margin and the iliac crest.
  Abdominal wall muscles (external oblique, internal oblique, and transversus abdominis) will be visualized.
  Bowel movement and visualization of hypoechoic peritoneum would further guide the block.
  The needle will be inserted in-plane and advanced until the tip is between the internal oblique and the transversus abdominis muscle.
  After negative aspiration, 20 mL of 0.25% bupivacaine is injected in a 5ml increment ,aspirating after every 5ml injection.
  Same procedure will be repeated on the other side.
  Other Names: TAP
  Arms: Transversus abdominis plane block

SUMMARY:
Hysterectomy is the second most common major Obstetric/gynecology procedure worldwide and one of the most common procedures in our institute. Post-operative pain is one of the most common complications following hysterectomy. Patients report moderate to severe pain following hysterectomy. Transversus abdominis plane block(TAP) is an established technique for abdominal and pelvic analgesia. Although efficient as an analgesic technique, it lacks visceral analgesia.Erector spinae plane block (ESP) is one of the newer developed regional techniques. Initially developed for Thoracic Neuropathic Pain by Forero et al, its use has expanded to include thoracic, abdominal and even femoral and below knee operative pain management.

Objective:

The objective of this study is to compare the ESP block with the TAP block for postoperative pain management in cases undergoing Total abdominal hysterectomy.

Methods:

A hospital based randomized, prospective, interventional study will be performed on all consenting patients undergoing total abdominal hysterectomy under general anesthesia. The required number of participants will be selected by probability sampling.

Fourty four female participants posted for elective Total abdominal hysterectomy under general anesthesia will be randomized onto two groups. The process of randomisation will be via computer generated randomization sequence.Each of the group will receive either of the two intervention after the completion of operative procedure. The post operative anelgesia duration and NRS score will be compared between the two groups.

Approval will be taken from the Institutional Review Committee (IRC) of Institute of Medicine.

Written consent will be taken prior to the data collection. Data will be entered in Microsoft Excel and errors will be checked. The clean data will be transferred into SPSS v 20 for analysis The results will be presented in terms of frequency percentage and table The associations will be established.

DETAILED DESCRIPTION:
Background

Hysterectomy is the second most common major Obstetric/gynecology procedure worldwide and one of the most common surgical procedure in our institute. Multiple indications like symptomatic uterine leiomyomas, abnormal uterine bleeding, endometriosis, and prolapse exist to warrant hysterectomy in a woman. By the age of 60, 1 in every 3 women in the US undergoes hysterectomy.

Multiple approaches and multiple techniques of hysterectomy exist.Approaches can be abdominal with pfannenstiel or low midline and Vaginal with paracervical incision. Techniques can be open, laparoscopic and even robot-assisted. The common approach in our resource limited setup is open abdominal with pfannenstiel incision.

Effective pain management plays a crucial role in reducing discomfort, aids in earlier mobilization, shortens hospital stay, reduces hospital cost, and increases patient satisfaction. The pain following hysterectomy is of moderate to severe grade. Many factors can influence post hysterectomy pain. Pre operative pain, extent of incision, approach to surgery, intra op and post operative pain management, age, socioeconomic status, presence of other painful sites all are risk factors for post hysterectomy pain. Adequate pain management is vital not only for patient comfort but also aids in early mobilization, improves functions, reduces venous thromboembolism risk and accelerates discharge. Furthermore in a Danish study by Birgitte Brandsborg using Danish Hysterectomy Database, the arthur noted the development of chronic Postoperative pain in 32% of all patients undergoing the procedure. One of the risk factors in the study was inadequate management of pain during preoperative and intraoperative periods.

Studies have shown pain perception in females to be higher than male population. Despite this women receive less pain management than men. Study by Esther H Chen et al on pain abdomen patients in the emergency department showed how women were less likely to get opioid analgesia, and had to wait longer to get analgesia to receive their dosing. All of these factors can play a significant role in increased pain and incidence of chronic pain in females.

Management of acute pain following surgery using a multimodal approach rather than a single narcotic/non-narcotic is recommended by the American Society of Anesthesiologists. Multimodal analgesia with focus on different sites of pain signals to prevent side effect of single medication is the current practice. It normally involves using various regional techniques, systemic and local medication. Regional techniques include epidural analgesia, local wound infiltration, TAP(Transversus abdominal plain) block, TENS(Transcutaneous Electrical Nerve Stimulation). Systemic medications include opioids, NSAIDs, Gabapentin, NMDA antagonists like Ketamine.

The Transversus abdominis plane(TAP) block is a regional injection of local anesthetic between the transversus abdominis and internal oblique muscle planes. TAP block affects the sensory nerves of the anterolateral abdominal wall (T6-L1) that innervate the abdomen. First described by Rafi as a single shot fascial analgesia technique at the lumbar triangle of petit.Local anesthetic is then injected between the internal oblique and transversus abdominis muscles. TAP block can also be applied with USG guidance. In a USG guided approach the probe is kept at the transverse plane between the lower costal margin and the iliac crest in the midaxillary line. Use of USG has made Transversus abdominis plane block relatively easy. The main disadvantage of TAP block is the lack of blockage of visceral pain. Visceral pain occurs when pain receptors in the pelvis, abdomen, chest, or intestines are activated. In a major surgery like TAH, blockage of somatic pain alone might not be enough.

Erector spinae plane block (ESP) is one of the newer developed regional techniques. Erector spinae (ES) consists of three columns of muscles: iliocostalis, longissimus, and spinalis. The three muscles run parallel to each other along the vertebra and extend from the lower back of the skull down to the pelvis. The erector spinae fascia extends from the nuchal fascia cranially to the sacrum caudally, local anesthetic agents extend through several levels, and the block can be effective over a large area. Initially developed for Thoracic Neuropathic Pain by Forero et al, its use has expanded to include thoracic, abdominal and even femoral and below knee operative pain management. The ESP block anesthetizes the ventral and dorsal rami of thoracic and lumbar nerves that give the sympathetic fibers. The technique involves injection of a local anesthetic in the plane between the erector spinae muscle and the spinal transverse processes. Dermatomes covered by ESP block depend on the point of entry, concentration, and the volume of local anesthetic used. The proposed advantages of this technique over the Transversus abdominis plane block are the increased duration of analgesia, presence of visceral block, easier administration and decreased side effect profile.

Kamel et al in 2020 compared bilateral ultrasound-guided Erector spinae Plane block against Transversus abdominis Plane Block. A total of 48 ASA PS 1 and 2 patients were randomly selected and grouped into ES and TA groups. Following TAH, the assigned procedure was done. Visual Analog Scale scores at 30 minutes, 2, 4, 6, 8, 12, 16, 20, and 24 hours post surgery were statistically significantly lower in the ES group compared with the TA group. The time required for the requirement of first morphine was statistically significantly prolonged in the ES group (14.81± 3.52 hours) compared with the TA group (10.58 ± 2.35 hours). The total amount of morphine consumption in 24 hours postoperatively was decreased in the ES group; P = 0.01. Incidence of postoperative nausea and vomiting was higher but statistically insignificant in the TA group than the ES group. There were statistically significant numbers of unsatisfied patients in the TA group compared with the ES group.

Kamel AAF, Amin OAI, Ibrahem MAM. Bilateral Ultrasound-Guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block on Postoperative Analgesia after Total Abdominal Hysterectomy. Pain Physician. 2020 Jul;23(4):375-382. PMID: 32709172.

Rationale of the study

Transversus Abdominis plane block is an established technique for abdominal and pelvic analgesia including post-operative pain management in Total abdominal hysterectomy.

Although efficient in controlling somatic pain, it doesnot provide complete analgesia. In cases of traction of peritoneum and handling of intraperitoneal organs, it is unable to provide visceral analgesia.

Erector spinae plane block is a newer technique proposed for pectoral, lumbar and abdominal procedures. The advantages of this technique over the Transversus abdominis plane block are the increased duration of analgesia, presence of visceral block, easier administration and decreased side effect profile. As such ESP block used in patients undergoing TAH might lead to better postoperative outcome for the patient.

General objective

To compare the ESP block with the TAP block for postoperative pain management in cases undergoing total abdominal hysterectomy

Specific objectives

Primary objective To compare the time of first rescue analgesia in ESP block group vs TAP block group To calculate and compare 24 hours of rescue analgesia consumption in ESP block group and TAP block group To measure and compare NRS score in ESP block and TAP block group at 0, 1, 6,8,12, 24hrs Secondary objective To determine and compare side effects-Respiratory depression, Sedation,motor block and complication of each modalities

Research hypothesis

Is ESP block better than TAP block for postoperative pain management in cases undergoing total abdominal hysterectomy? Research hypothesis Null hypothesis (H0): ESP block is not superior to TAP block for postoperative pain management in case undergoing total abdominal hysterectomy Alternative hypothesis (H1): ESP block is superior to TAP block for postoperative pain management in case undergoing total abdominal hysterectomy Expected outcome H0 ≠ H1

Sample size calculation

Sample size was derived based on comparative study on ESP block and TAP block by Kamel et al.

za=1.96 at 95% confidence level zβ=1.65 at 95% power using formula n=2(za+zβ )2 S2d2 Mean time for requirement of first morphine dose in ESP group= 14.81 hours , SD= 3.52, mean in TAP group = 10.58 hours , SD= 2.35 d= mean difference = 14.81 - 10.58 = 4.23 S = 3.52 (larger among 2 groups) size is n= 19 per group Considering 10% dropout, an addition of 2 in each group is warranted. Final n=22 per group

Randomization And Blinding

Computer controlled randomization via Microsoft Excel version 2010 Patients will be allocated to either of the two groups. Group A /ESP block Group B /TAP block Allocation concealment via sealed envelope method Blinding- The envelopes will be opened by an attending nurse not involved in the study before completion of the operation .

The study drug will be prepared by the anesthesiologist who will perform the block The data will be filled by another anesthesiologist/medical officer not involved in the block.

Management protocol of participants

One day prior to Operative procedure Pre anesthetic check up will be done in the ward. Patients will be explained about the purpose of the study, the possible benefits, and any risks of the procedure.

Patients will be taught about Numerical Rating Score(NRS). Written informed consent will be obtained from all participants.

In the operating room Intravenous access will be established. All ASA standard I and II monitors will be connected. Baseline vitals will be monitored and recorded. All patients will be subjected to a standardized anesthetic protocol. General Anesthesia will be induced with Inj Fentanyl 2mcg/kg and dosing would be recorded. Inj Propofol in titrating dose Any additional dosing of analgesia given during induction will be documented. Neuromuscular blockade used for endotracheal intubation will be either Vecuronium 0.1mg/kg or Rocuronium 1 mg/kg.

Ventilation parameter as per standard anesthetic practice in our institute. Maintenance of anesthesia will be done with Isoflurane (1% to 2%) and oxygen. Ringer lactate solution will be infused throughout the surgery as per standard practice in our institute.

Analgesia during the perioperative period will be standardized Inj Paracetamol 15 mg/kg infusion post induction Inj Fentanyl 0.5mcg/kg per hour of perioperative period and any additional dosing of analgesia will be recorded.

PONV prophylaxis will be standardized in both groups of patient Inj Dexamethasone 4mg single dose immediate post induction Inj Ondansatran 4mg single dose 15 to 20 minutes before extubation.

Before completion of the operation:

Sealed envelope will be opened by the nursing staff not involved in the study. The patient will be grouped as Group A (ESP block) Group B (TAP block) Two syringes of 20 ml 0.25% concentration Bupivacaine will be prepared by the attending anesthesiologist.

Patient will be positioned in the lateral position in the ESP block group and will be kept in supine position for the TAP block group.

Under all antiseptic precautions, the USG guided bilateral ESP block/TAP block will be given by an attending anesthesiologist.

Maintenance of anesthesia with isoflurane and oxygen will be continued throughout the block.

Anesthetic gas will be switched off following the block. Patient will be extubated as per standard anesthetic protocol. Patient will be transferred to the recovery room. Patients will be held in recovery ward/PACU until adequate recovery from anesthesia as judged by the Modified Aldrete score. Score ≥ 9 will be deemed adequate.

Post-operative pain assessment will be done with Numeric Rating Scale(NRS). NRS is accessed at 0,1,6,8,12,24 hours by nursing staff. The time 0 would be the first assessment of pain done in the postoperative recovery unit of our operating theater.

Data management and statistical analysis

Statistical analysis will be done after completion of the study. The collected data will be entered into the Microsoft Excel sheet and will be exported to the Statistical Package for Social Sciences, version 25 for analysis.

Demographic data (age, weight, height, BMI) will be expressed as mean or median and standard deviation and range, as appropriate.

Duration of rescue analgesia, doses, and NRS scores will be expressed as mean and standard deviation and compared using independent sample t-test Qualitative data will be expressed as number and percentage and will be analyzed by the chi-square test The data will be subsequently analyzed; a p-value of <0.05 will be considered significant with 95% confidence limit.

Limitations of the study

Post operative pain or any pain are subjective experiences. It can be difficult to quantify and compare various outcomes.

Due to the nature of the study patient cannot be truly blinded as the site of block are further apart.

Safety considerations

Both ESP and TAP blocks are relatively safe analgesia techniques. Calculated dosing based on weight of the patient lowers the incidence of local anesthetic toxicity.

The use of USG and injecting local anesthesia guided by intrafascial movement of local anesthesia make them safer.

Follow up of vitals and side effect profiles of each group also improve their safety profile. Patient will be continually monitored postoperatively for 24hrs.

Ethical issues

The study will only commence after approval from Institutional Review Committee,IOM and NHRC.

It will be registered in the Nepal Clinical Trials Registry of the Nepal Health Research Council before enrollment.

This study will be reviewed continuously by guide, coguide and the MMC Anesthesiology department.

The participants involved in the research project will be volunteers and informed participants.

Written informed consent will be obtained from all the participant included in the study.

The participants will be given the right to abstain from participation in the study or to withdraw consent to participate at any time of the study without reprisal.

Every precaution will be taken to respect the privacy of the participants , the confidentiality of the participants' information and to minimize the impact of the study on participants physical and mental integrity and personality.

Data recorded from the participants will be encrypted and stored in TUTH Anesthesiology department computer. The excel sheet in which data of the participants is recorded will be password protected.

Data recorded from participants will not be shared with any third party. The intervention performing in this research are standard practice of anaesthesia in our institute.

ELIGIBILITY:
Inclusion Criteria:

* All cases undergoing total abdominal hysterectomy under GA
* Age >18 years
* Elective cases
* ASA PS I & II

Exclusion Criteria:

* Patient refusal
* Patient with contraindication to peripheral Nerve blocks
* Allergy to local anesthetics
* Weight less than 50kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Time of first rescue analgesia within 24hours | 24hours
  Rescue analgesia used injection Tramadol, given if Numerical rating score(NRS) >3 withing 24hours of the procedure.

SECONDARY OUTCOMES:
Total amount of rescue analgesia. | 24hours
  Amount of rescue analgesia(inj tramadol) given to the patient withing 24hours of the procedure.
Pain assessment at set time | 24hours
  Pain assessment done with Numerical rating score(0-10) at 0,1,6,8,12,24 hours. Numerical Rating score of 0 represents 'no pain at all' whereas 10 represents 'the worst pain ever possible'
Comparision of side effect: Incidence of Respiratory depression,Incidence of sedation, motor block, postoperative nausea and vomiting postoperative nausea and vomiting of intervention | 24hours
  The number of episodes of Respiratory depression, sedation, motor block, postoperative nausea and vomiting with each intervention will be recorded.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Wechter ME, Geller EJ, Nguyen TV, Visco AG. Hysterectomy rates in the United States, 2003. Obstet Gynecol. 2007 Nov;110(5):1091-5. doi: 10.1097/01.AOG.0000285997.38553.4b. PMID 17978124
- [Background] Lissauer J, Mancuso K, Merritt C, Prabhakar A, Kaye AD, Urman RD. Evolution of the transversus abdominis plane block and its role in postoperative analgesia. Best Pract Res Clin Anaesthesiol. 2014 Jun;28(2):117-26. doi: 10.1016/j.bpa.2014.04.001. Epub 2014 May 9. PMID 24993433
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kamel AAF, Amin OAI, Ibrahem MAM. Bilateral Ultrasound-Guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block on Postoperative Analgesia after Total Abdominal Hysterectomy. Pain Physician. 2020 Jul;23(4):375-382. PMID 32709172
- [Background] Balaban O, Aydin T. Lumbar erector spinae plane catheterization for continuous postoperative analgesia in total knee arthroplasty: A case report. J Clin Anesth. 2019 Aug;55:138-139. doi: 10.1016/j.jclinane.2018.12.017. Epub 2019 Jan 15. No abstract available. PMID 30658328
- [Background] Sinatra R. Causes and consequences of inadequate management of acute pain. Pain Med. 2010 Dec;11(12):1859-71. doi: 10.1111/j.1526-4637.2010.00983.x. Epub 2010 Oct 28. PMID 21040438
- [Background] Pieretti S, Di Giannuario A, Di Giovannandrea R, Marzoli F, Piccaro G, Minosi P, Aloisi AM. Gender differences in pain and its relief. Ann Ist Super Sanita. 2016 Apr-Jun;52(2):184-9. doi: 10.4415/ANN_16_02_09. PMID 27364392
- [Background] Chen EH, Shofer FS, Dean AJ, Hollander JE, Baxt WG, Robey JL, Sease KL, Mills AM. Gender disparity in analgesic treatment of emergency department patients with acute abdominal pain. Acad Emerg Med. 2008 May;15(5):414-8. doi: 10.1111/j.1553-2712.2008.00100.x. PMID 18439195
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Boules ML, Goda AS, Abdelhady MA, Abu El-Nour Abd El-Azeem SA, Hamed MA. Comparison of Analgesic Effect Between Erector Spinae Plane Block and Transversus Abdominis Plane Block After Elective Cesarean Section: A Prospective Randomized Single-Blind Controlled Study. J Pain Res. 2020 May 19;13:1073-1080. doi: 10.2147/JPR.S253343. eCollection 2020. PMID 32547172
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Hamed MA, Goda AS, Basiony MM, Fargaly OS, Abdelhady MA. Erector spinae plane block for postoperative analgesia in patients undergoing total abdominal hysterectomy: a randomized controlled study original study. J Pain Res. 2019 Apr 30;12:1393-1398. doi: 10.2147/JPR.S196501. eCollection 2019. PMID 31118757
- [Background] Altinpulluk EY, Ozdilek A, Colakoglu N, Beyoglu CA, Ertas A, Uzel M, Yildirim FG, Altindas F. Bilateral postoperative ultrasound-guided erector spinae plane block in open abdominal hysterectomy: a case series and cadaveric investigation. Rom J Anaesth Intensive Care. 2019 Apr;26(1):83-88. doi: 10.2478/rjaic-2019-0013. PMID 31111101
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158

DOCUMENTS (1):
  • Informed Consent Form (2022-08-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT05521841/ICF_000.pdf